CLINICAL TRIAL: NCT07289178
Title: Effect of Liposome Bupivacaine Serratus Plane Block on Postoperative Hyperalgesia and Chronic Post-surgical Pain in Patients Undergoing Radical Mastectomy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Haixia Jiang, Clinical Professor of The first affiliated hospital of KUNMING medical university, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1stKunmingMC2
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Serratus Plane Block; Postoperative Hyperalgesia; Chronic Post-surgical Pain; Liposomal Bupivacaine; Radical Mastectomy Surgery
Keywords: serratus plane block; postoperative hyperalgesia; chronic post-surgical pain; Liposomal Bupivacaine; Radical mastectomy surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-dose remifentanil saline serratus plane block group (Placebo Comparator): Anesthesia induction began with continuous infusion of remifentanil until skin suturing was completed at a low dose of 0.1 μg/(kg·min). After anesthesia induction, 20 ml of normal saline was used for the preoperative quadratus lumborum block group.
  Interventions: Procedure: Serratus Plane block (single injection)
- Hight-dose remifentanil saline serratus plane block group (Placebo Comparator): Anesthesia induction began with continuous infusion of remifentanil until skin suturing was completed at a high dose of remifentanil 0.3 μg/(kg·min). After anesthesia induction, 20 ml of normal saline was used for the preoperative serratus anterior muscle block group.
  Interventions: Procedure: Serratus Plane block (single injection)
- Highight-dose remifentanil with 0.375% ropivacaine serratus plane block group (Active Comparator): Anesthesia induction began with continuous infusion of remifentanil until the completion of skin suturing, with a high-dose remifentanil infusion rate of 0.3 μg/(kg·min). After anesthesia induction, a pre-saw muscle block was performed using 20 ml of 0.375% ropivacaine.
  Interventions: Procedure: Serratus Plane block (single injection)
- Highight-dose remifentanil with 0.665% Liposomal Bupivacaine serratus plane block group (Experimental): Anesthesia induction began with a continuous infusion of remifentanil until the end of skin suturing, at a high dose of remifentanil infusion at 0.3 μg/(kg·min). After anesthesia induction, 20 ml of 0.665% liposomal bupivacaine was administered for a serratus plane block
  Interventions: Procedure: Serratus Plane block (single injection)

INTERVENTIONS:
Procedure: Serratus Plane block (single injection) — After anesthesia induction, the same experienced anesthesiologist performed an ultrasound-guided serratus anterior plane block on the surgical side. The skin was routinely disinfected and draped. A linear 10-13 MHz ultrasound probe was used to locate the 5th rib along the mid-axillary line to identify the superficial latissimus dorsi and the deep serratus anterior muscles. A 22G (80 mm) nerve block needle was inserted in-plane from anterolateral to posteroinferior. When the needle tip reached the surface of the serratus anterior muscle, with clear visualization of the tip in place, no aspiration of fluid, and no air, a test dose of 2 ml was first administered. After a hypoechoic area was observed on the ultrasound, and no blood or air was aspirated again, 20 ml of 0.375% ropivacaine was slowly injected in the ropivacaine group, 20 ml of 0.665% liposomal bupivacaine in the liposomal bupivacaine group, and 20 ml of saline in the placebo group, with real-time ultrasound visualization of t

SUMMARY:
Radical mastectomy is currently the mainstream surgical treatment for breast cancer. Patients often experience significant postoperative pain, and some may develop chronic pain. General anesthesia is commonly used, with remifentanil being the most frequently used intraoperative analgesic. However, prolonged high-dose use of remifentanil can induce opioid-induced hyperalgesia (OIH). Previous studies have shown that serratus anterior plane block can reduce acute postoperative pain after radical mastectomy, but it remains unclear whether it can reduce postoperative pain sensitization and the incidence of chronic pain. Liposomal bupivacaine is a new long-acting local anesthetic with an effect lasting up to 72 hours. This study aims to investigate the effect of liposomal bupivacaine serratus anterior plane block on postoperative pain sensitization and chronic pain in patients undergoing radical mastectomy, providing a reference for clinical treatment. The study includes 120 participants. A tactile measurement kit is used to measure the mechanical pain threshold around the surgical incision preoperatively and at 24 and 48 hours postoperatively, as well as postoperative persistent pain scores at 7 days, 1 month, 3 months, and 6 months. The data will then be analyzed to draw conclusions.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind trial. Approved by the hospital ethics committee, patients signed informed consent forms. A total of 120 patients scheduled for elective radical mastectomy under general anesthesia were selected, with ASA classifications I-IV, aged 18-80 years, and BMI <30 kg/m². They were randomly divided into four groups using a computer-generated randomization method: low-dose remifentanil with saline pre-pectoral nerve block group (LR NS), high-dose remifentanil with saline pre-pectoral nerve block group (HR NS), high-dose remifentanil with ropivacaine pre-pectoral nerve block group (HR L), and high-dose remifentanil with liposomal bupivacaine pre-pectoral nerve block group (HR B). Patient general information, anesthesia time, surgery time, remifentanil dosage, and the doses of saline, ropivacaine, and liposomal bupivacaine for the pre-pectoral nerve block were recorded. Non-invasive blood pressure (MAP) and heart rate (HR) were measured before anesthesia induction, before intubation, immediately after intubation, at skin incision, during skin closure, and at extubation. Intraoperative vasoactive drugs usage and doses were also recorded. Postoperative NRS pain scores were assessed at 1h, 6h, 24h, and 48h, along with the amount of rescue analgesics used within 24h after surgery, the number of patients requiring rescue analgesia, and any adverse reactions such as postoperative nausea, vomiting, dizziness, drowsiness, and respiratory depression. Preoperatively and at 24h and 48h postoperatively, patients' mechanical pain thresholds around the surgical incision area and forearm were measured using a tactile measurement kit (Von Frey filaments). Postoperative recovery quality scores were recorded on day 1 and day 3, and persistent postoperative pain assessment scores were recorded at 7 days, 1 month, 3 months, and 6 months after surgery.

The research solutions, including remifentanil (40 μg/mL), 0.665% bupivacaine liposome (20 mL), and 0.375% ropivacaine (20 mL), were prepared by specialized anesthesiologists. The placebo group was prepared with only normal saline, and the preparation process was kept confidential from the investigators. Anesthesia was administered by two designated anesthesiologists according to the established trial protocol. No premedication was given to any patient. Upon entering the operating room, heart rate (HR), standard electrocardiogram (ECG), oxygen saturation (SpO2), and non-invasive blood pressure (MAP) were monitored every 5 minutes. The mean of three consecutive HR and MAP values was taken as the baseline. Bispectral index (BIS) and neuromuscular monitoring with 4-train-of-four (TOF) stimuli were also conducted. In the low-dose remifentanil group (LR), remifentanil was infused at 0.1 μg/(kg·min); in the high-dose remifentanil group (HR), remifentanil was continuously infused at 0.3 μg/(kg·min). During induction of anesthesia, remifentanil infusion continued until the completion of skin closure. General anesthesia was induced with propofol 2.0 mg/kg and rocuronium 0.9 mg/kg. When BIS < 60 and TOF count was 0, an enhanced endotracheal tube was inserted orally using either a direct laryngoscope or a video laryngoscope, using a size 7.0 tube for female patients. Mechanical ventilation was controlled, with fresh gas flow of oxygen-air mixture (50% O2) at 2 L/min, tidal volume 6-8 mL/kg, and respiratory rate of 10-12 breaths/min, maintaining end-tidal CO2 at 35-40 mmHg. Anesthesia was maintained with sevoflurane to keep BIS between 40-60. Rocuronium 0.2 mg/kg was administered intermittently if the TOF count reached 0.4. When mean arterial pressure < 60 mmHg, 6 mg of ephedrine was given intravenously. If heart rate < 50 bpm, 0.5 mg of atropine was given intravenously. At the end of skin closure, sevoflurane and remifentanil infusion were stopped, and 50 mg of flurbiprofen ester was administered intravenously for analgesia. Once the TOF ratio recovered to greater than 90%, 2 mg/kg of sugammadex sodium was given to reverse residual neuromuscular blockade. The endotracheal tube was removed when the patient had sufficient spontaneous tidal volume and was awake enough to respond correctly to verbal commands, and the patient was transferred to the PACU. When the Steward score reached 6, the patient was transferred to the ward.

After anesthesia induction, the same experienced anesthesiologist performed an ultrasound-guided serratus anterior plane block on the surgical side. The skin was routinely disinfected and draped. A linear 10-13 MHz ultrasound probe was used to locate the 5th rib along the mid-axillary line to identify the superficial latissimus dorsi and the deep serratus anterior muscles. A 22G (80 mm) nerve block needle was inserted in-plane from anterolateral to posteroinferior. When the needle tip reached the surface of the serratus anterior muscle, with clear visualization of the tip in place, no aspiration of fluid, and no air, a test dose of 2 ml was first administered. After a hypoechoic area was observed on the ultrasound, and no blood or air was aspirated again, 20 ml of 0.375% ropivacaine was slowly injected in the ropivacaine group, 20 ml of 0.665% liposomal bupivacaine in the liposomal bupivacaine group, and 20 ml of saline in the placebo group, with real-time ultrasound visualization of the spread of the local anesthetic (or saline). Throughout the procedure, the patient's vital signs were monitored. In case of local anesthetic toxicity, basic life support was immediately initiated, 20% lipid emulsion was rapidly administered intravenously, and preparations were made for prolonged monitoring and advanced life support.

Tactile measurement kits (Von Frey filaments) were used to assess the mechanical pain sensitivity thresholds of patients around the surgical incision and on the forearm at preoperative (T1), 24 hours postoperative (T2), and 48 hours postoperative (T3) time points. The method for measuring mechanical pain thresholds around the incision involved testing at points 2 cm from both ends of the surgical incision and 2 cm below the center of the incision, and the average of the three measurements was taken. For the forearm, measurements were taken at points 3, 6, and 9 cm from the midpoint of the elbow, and again, the average of the three points was calculated. The tactile measurement kit consists of filaments of varying thickness, with filament weight corresponding to different levels of mechanical stimulation intensity. The specific measurement procedure was as follows: the patient closed their eyes, and the investigator applied the filaments vertically to the patient's skin until the filament bent, holding for 1.5 seconds; filaments ranging from 15 to 180 g were used, starting with the 15 g filament and progressing in ascending order; if the patient showed no response or reported sensation as touch, the filament strength was increased; if the patient reported a tingling sensation, the filament strength was decreased. The up-down method was used to calculate the mechanical pain threshold. The up-down method is a classical approach to measure mechanical pain thresholds and estimates the 50% mechanical pain threshold, calculated using the formula 50% threshold (g) = Xf + kd, where Xf represents the weight corresponding to the last filament stimulus, k is the maximum likelihood estimation value, and d is the log value of the difference between consecutive stimulus intensities. A smaller calculated value indicates a lower pain threshold.

Patients were assessed for persistent pain at 7 days, 1 month, 3 months, and 6 months postoperatively. The evaluation questions included: (1) Whether chronic pain exists;(2) Type of pain: stabbing pain, electric shock-like pain, swelling pain, numbness of the skin, etc.;(3) Pain location: breast area, ipsilateral axilla, ipsilateral upper arm, other areas (such as lower back pain and headache). Pain intensity was assessed using the NRS from 0 to 10. Pain levels were calculated separately at rest (for example, pain intensity when sitting or lying down) and during movement (for example, pain intensity when moving the ipsilateral upper arm or walking);(4) Whether pain changed after adjuvant therapy: post-operative adjuvant therapy includes radiotherapy, chemotherapy, endocrine therapy, or HER2-targeted therapy;(5) Whether pain was treated: taking analgesics, acupuncture, electrotherapy, and nerve blocks;(6) Whether the patient had previous surgeries and whether they also had long-term pain symptoms.

Statistical analyses were performed using SPSS 17.0 software. The Shapiro-Wilk test was used to assess the normality of data in each group. Normally distributed measurement data were expressed as mean ± standard deviation and analyzed using one-way or repeated measures ANOVA, with Bonferroni test for pairwise comparisons. Non-normally distributed measurement data were expressed as median (M) and interquartile range (IQR) and analyzed using the non-parametric Kruskal-Wallis test, with Mann-Whitney U test for pairwise comparisons. Categorical data were compared using the χ2 test or Fisher's exact test. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Select patients scheduled for elective radical mastectomy for breast cancer under general anesthesia, ASA grade I-IV, aged 18-80 years.

Exclusion Criteria:

Allergy to the anesthetics used, infection at the puncture site, history of chronic pain and current use of opioid analgesics, history of chest surgery or trauma, drug or alcohol dependence, neurological or psychiatric disorders, severe hepatic or renal insufficiency, pregnancy, body mass index (BMI) greater than 30 kg/m².

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical pain threshold around the postoperative incision | Detected preoperatively (T1), 24 hours postoperatively (T2), and 48 hours postoperatively (T3)
  Tactile measurement kits (Von Frey filaments) were used to assess patients' mechanical pain detection thresholds around the surgical incision area and the forearm preoperatively (T1), 24 hours postoperatively (T2), and 48 hours postoperatively (T3). The method for measuring mechanical pain thresholds involved measuring the threshold around the incision at two points 2 cm from either end of the incision and one point 2 cm below the middle of the incision, with the average of the three points taken as the final value. For the forearm, measurements were taken at points 3, 6, and 9 cm from the midpoint of the elbow, and the average of these three points was calculated similarly. The tactile measurement kit consists of filaments of varying thicknesses, with the filament weight corresponding to different levels of mechanical stimulus intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China